CLINICAL TRIAL: NCT02992353
Title: Single-port Versus Two-port Versus Three-port Video Assisted Thoracoscopic Pulmonary Resection on Non-small Cell Lung Cancer: a Prospective Randomised Controlled Trial
Brief Title: Single-port, Two-port Versus Three-port VATS on Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ju-Wei Mu, MD, PHD, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z161100000116044
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Lung Neoplasm
Keywords: VATS; NSCLC; recurrence rate
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Three-port pulmonary resection surgery (Active Comparator): Treated by traditional video assisted thoracoscopic three-port pulmonary resection in the centers with enough experience in VATS and the volume ≧50 cases each year.
  Interventions: Procedure: Three-port pulmonary resection surgery
- Single-port or two-port surgery (Active Comparator): Treated by minimally invasive video assisted thoracoscopic single-port or two-port pulmonary resection in the centers with enough experience in VATS and the volume ≧50 cases each year.
  Interventions: Procedure: Single-port or two-port surgery

INTERVENTIONS:
Procedure: Three-port pulmonary resection surgery — Three-port pulmonary resection surgery
  Arms: Three-port pulmonary resection surgery
Procedure: Single-port or two-port surgery — Single-port or two-port pulmonary resection surgery
  Arms: Single-port or two-port surgery

SUMMARY:
In china, the incidence and death rate of lung cancer is 48.32 per 100 000 person-years and 39.27 per 100 000 person-years, respectively, the highest in malignant tumor. Surgical operation is still main treatment means to resectable NSCLC. VATS pulmonary resection is performed in clinical operation with the aim of decreasing postoperative complications morbidity. The mechanisms may be due to minimize the inflammation reaction to surgical injury. There are some trials regarding two-port VATS versus three-port VATS versus four-port VATS or single-port VATS versus three-port VATS. However, there is no prospective randomised controlled trial regarding Single-port versus two-port versus three-port video assisted thoracoscopic pulmonary resection on NSCLC. So, we hope to demonstrate that single-port and two-port VATS were feasible and safe through the trial, and we hope the results of our study will provide a high level of clinical evidence for choosing the best operative approach in VATS.

DETAILED DESCRIPTION:
Introduction: In china, the incidence and death rate of lung cancer is 48.32 per 100 000 person-years and 39.27 per 100 000 person-years, respectively, the highest in malignant tumor. Surgical operation is still main treatment means to resectable NSCLC. VATS pulmonary resection is performed in clinical operation with the aim of decreasing postoperative complications morbidity. The mechanisms may be due to minimize the inflammation reaction to surgical injury. There are some trials regarding two-port VATS versus three-port VATS versus four-port VATS or single-port VATS versus three-port VATS. However, there is no prospective randomised controlled trial regarding Single-port versus two-port versus three-port video assisted thoracoscopic pulmonary resection on NSCLC. So, we hope to demonstrate that single-port and two-port VATS were feasible and safe through the trial, and we hope the results of our study will provide a high level of clinical evidence for choosing the best operative approach in VATS.

Methods and analysis: this is a three years prospective randomised controlled trial, which aims to attest the safety and feasibility of simple-port VATS and two-port VATS. Group A, B and C receives single-port VATS, two-port VATS and three-port VATS pulmonary resection respectively. The primary endpoint is postoperative recurrence rate. The secondary endpoints include other postoperative complications morbidity , such as the number and location of lymph nodes dissected、operation time, intraoperative volume of blood loss, hospital stays, hospitalization expenses, quantity of using antalgica, change of pulmonary function. 70 patients are enrolled per group in three years, after adding 10% loss of the sample, 77 patients will be required for each group so a total of 231 patients will be enrolled into the study in the end.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years;
* cT1-3N0-1M0 diagnosed by chest CT or PET-CT before operation;
* ECOG PS scores≤2;
* The patients sign informed consents by themselves.

Exclusion Criteria:

* Inability to tolerance of tracheal intubation and general anesthesia;
* ECOG PS scores>2;
* Severe comorbidities including: Angina occurs in 3 months, uncontrolled hypertension, Congestive heart failure, a history of myocardial infarction in 6 months before admission, severe arrhythmia, severe liver, kidney or other metabolic diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Local recurrence | 2 years
  two-year local recurrence rate after surgery

SECONDARY OUTCOMES:
Postoperative respiratory complications | 30 days after surgery
  Systematic Classification of Morbidity and Mortality After Thoracic Surgery. Grade I, any complication without need for pharmacologic treatment or other intervention. Grade II, any complication that requires pharmacologic treatment or minor intervention only. Grade III , any complication that requires surgical, radiologic, endoscopic intervention, or multitherapy.
  Grade IV, any complication requiring intensive care unit management and life support.
  Grade V, any complication leading to the death of the patient.
Lymph node dissection | Intraoperation
  During the surgery, lymph node dissection were performed. The number of removed lymph-nodes were recorded according to the postoperative pathological diagnosis, and the stations of the lymph node were recorded according to the International Association for the Study of Lung Cancer (IASLC) Lymph Node Map.
Blood loss | Intraoperation
  blood loss during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Juwei Mu, MD, Principal Investigator — Beijing Municipal Science & Technology Commission
Locations (1):
- Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided